CLINICAL TRIAL: NCT01787448
Title: Repeat-insult Patch Test (Ript) of Ibuprofen 5% Topical Gel in Human Volunteers
Brief Title: RIPT of Ibuprofen Topical Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B3491007
Record Dates: First submitted 2012-12-05; First posted 2013-02-08 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: repeat insult patch test
MeSH Terms: conditions — Pain | interventions — Gels; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen 5% topical gel (Experimental)
  Interventions: Drug: Topical gel vehicle
- Topical gel vehicle (Experimental)
  Interventions: Drug: Topical gel vehicle
- Sodium lauryl sulfate 0.1% (Active Comparator)
  Interventions: Drug: Sodium lauryl sulfate 0.1%
- Sodium chloride solution 0.9% (saline) (Sham Comparator)
  Interventions: Drug: Sodium chloride solution 0.9% (saline)

INTERVENTIONS:
Drug: Topical gel vehicle — 0.2 ml applied every 2 days (or 3 days if over the weekend) over 22 days (9 applications) followed by 10-14 day rest period and one subsequent re-application
  Arms: Ibuprofen 5% topical gel
Drug: Topical gel vehicle — 0.2 ml applied every 2 days (or 3 days if over the weekend) over 22 days (9 applications) followed by 10-14 day rest period and one subsequent re-application
  Arms: Topical gel vehicle
Drug: Sodium lauryl sulfate 0.1% — 0.2 ml applied every 2 days (or 3 days if over the weekend) over 22 days (9 applications) followed by 10-14 day rest period and one subsequent re-application
  Arms: Sodium lauryl sulfate 0.1%
Drug: Sodium chloride solution 0.9% (saline) — 0.2 ml applied every 2 days (or 3 days if over the weekend) over 22 days (9 applications) followed by 10-14 day rest period and one subsequent re-application
  Arms: Sodium chloride solution 0.9% (saline)

SUMMARY:
This study is being conducted to determine the potential of Ibuprofen 5% Topical Gel and its vehicle gel to cause sensitization after repeated topical application to healthy skin of human subjects under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female subjects 18 years of age or older, female subjects of childbearing potential and males are using an acceptable form of birth control, subjects are free of any systemic or dermatologic disorder

Exclusion Criteria:

Have any visible skin disease at the application site, not willing to stop use of systemic or topical analgesics, corticosteroids, or antihistamines, not willing to stop use of sunscreens, creams, or similar products on the back during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Dermal sensitization potential | 24-72 hours after last patch removal

SECONDARY OUTCOMES:
Cumulative Irritancy | 48-72 hours after each patch application
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | During study through 28 days after last product application

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Carlstadt, New Jersey, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491007&StudyName=RIPT%20of%20ibuprofen%20topical%20gel